CLINICAL TRIAL: NCT03642483
Title: Evaluation of an Early Screener to Identify Long-term Problems With Regard to Metabolic Control and Treatment Adherence Among Children and Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00374-G1
Record Dates: First submitted 2018-07-03; First posted 2018-08-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; metabolic control; psychosocial risk factors; FEPB; children; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Type 1 diabetes is one of the most common chronic illnesses among children and adolescents. Although, intensive medical care is provided for these patients, some of them have poor metabolic control. For example, only 21% of adolescents with type 1 diabetes in the USA achieve the recommended average blood sugar concentration (HbA1c<7.5%). This is a major problem, since chronic hyperglycemia is the primary cause of morbidity and mortality in type 1 diabetes and causes several serious complications, for example kidney failure, blindness, and stroke. Therefore, the International Society for Pediatric and Adolescent Diabetes (ISPAD) declared psychosocial factors, to be the most important risk factors of poor type 1 diabetes Management. Therefore, an instrument is needed to identify children and adolescents with poor metabolic control in their course of disease as soon as possible. With an early identification of such risk patients, better support can be provided. However, there is no such instrument yet for pediatric patients with type 1 diabetes. To fill this gap, a questionnaire (FEPB) based on the PAT 2.0© (Psychosocial Assessment Tool; an instrument used in oncology) was developed for this project.

Aim: The aim of this project is to evaluate and validate a new instrument (FEPB) for an early identification of children and adolescents with poor metabolic control in their course of disease in a longitudinal design.

Method: The sample consists of children and adolescents (age: 5-18 years), who were newly diagnosed with type 1 diabetes (2-4 weeks ago), and who are in care at the University Children's Hospital of Zurich. Structured interviews are conducted with the patients and the parents are asked to fill out some questionnaires at two times: first, 2-4 weeks after the diagnosis (T1) and second 6 month later (T2). With the new instrument (FEPB) a risk score can be calculated for each patient at T1. Statistical analysis will be performed to determine whether that risk score can predict which patients have poor metabolic control (HbA1c > 7.5%) at T2.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 Diabetes 2-4 weeks ago
* in care at the University Children's Hospital of Zurich
* German speaking

Exclusion Criteria:

* other severe illness that affects the diabetes Management
* severe developmental disorder
* pregnancy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic - University Children's Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
HbA1c | 10 minutes
  Glycated hemoglobin

SECONDARY OUTCOMES:
health-related quality of life (Chronic generic measure) | 5 minutes
  Assessed by questionnaire: DISABKIDS Chronic generic measure - short version (DCGM-12; the European DISABKIDS Group, 2012).
  Total score range: 12-60. The higher the score, the higher the health-related quality of life.
health-related quality of life (diabetes module) | 5 minutes
  Assessed by questionnaire: DISABKIDS diabetes module (The European DISABKIDS Group, 2012).
  Total score range: 10-50. The higher the score, the higher the health-related quality of life.
psychological health (Depression) | 10 minutes
  Assessed by questionnaire: German Version of the Children's Depression Inventory (Depressionsinventar für Kinder und Jugendliche [DIKJ]; Stiensmeier-Pelster, Braune-Krickau, Schürmann & Duda, 2014).
  Total score range: 0-58. The higher the score, the more depressed the participants are.
psychological health (Trait-Anxiety) | 5 minutes
  Assessed by questionnaire: German Version of the Trait-Anxiety Inventory for Children (Trait Angstinventar für Kinder [STAIK-T]; Unnewehr, Joormann, Schneider & Margraf, 1992).
  Total score range: 20-60. The higher the score, the higher the trait anxiety.
psychological health (Child Behavior) | 10 minutes
  Assessed by questionnaire: German Version of the Child Behavior Checklist (CBCL 6-18R; Döpfner, Plück & Kinnen, 2014) Total score range: 0-224. The higher the score, the more behavioral problems.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Landolt, Prof. dr., Principal Investigator — University Children's Hospital, Zurich; Daniel Konrad, Prof. dr., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Datye KA, Moore DJ, Russell WE, Jaser SS. A review of adolescent adherence in type 1 diabetes and the untapped potential of diabetes providers to improve outcomes. Curr Diab Rep. 2015 Aug;15(8):51. doi: 10.1007/s11892-015-0621-6. PMID 26084580
- [Background] Delamater AM. Psychological care of children and adolescents with diabetes. Pediatr Diabetes. 2009 Sep;10 Suppl 12:175-84. doi: 10.1111/j.1399-5448.2009.00580.x. No abstract available. PMID 19754628
- [Background] Kazak AE, Brier M, Alderfer MA, Reilly A, Fooks Parker S, Rogerwick S, Ditaranto S, Barakat LP. Screening for psychosocial risk in pediatric cancer. Pediatr Blood Cancer. 2012 Nov;59(5):822-7. doi: 10.1002/pbc.24166. Epub 2012 Apr 10. PMID 22492662
- [Background] Litmanovitch E, Geva R, Rachmiel M. Short and long term neuro-behavioral alterations in type 1 diabetes mellitus pediatric population. World J Diabetes. 2015 Mar 15;6(2):259-70. doi: 10.4239/wjd.v6.i2.259. PMID 25789107